CLINICAL TRIAL: NCT03890107
Title: Clinical Evaluation of a New Middle Ear Diagnostic to Support FDA Regulatory Clearance
Brief Title: Clinical Evaluation of the OtoSight
Status: Completed | Type: Observational
Sponsor: PhotoniCare, Inc. (Industry)
Collaborators: Carle Foundation Hospital (Other); Children's National Research Institute (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 000001; R44DC014599 (NIH)
Record Dates: First submitted 2019-03-18; First posted 2019-03-26 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Otitis Media
Keywords: Ear Infection; Ear tubes; Myringotomy; Otitis Media; Tympanostomy
MeSH Terms: conditions — Otitis Media; Otitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Middle ear effusion, if present
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Pediatric tympanostomy tube patients: Patients diagnosed with otitis media and scheduled for tympanostomy tube placement will be imaged with the OtoSight
  Interventions: Device: OtoSight Middle Ear Scope

INTERVENTIONS:
Device: OtoSight Middle Ear Scope — OtoSight imaging using a near-infrared laser

SUMMARY:
The objective of this study is to evaluate the imaging capabilities and image analysis performance of the OtoSight Middle Ear Scope in pediatric patients undergoing tympanostomy tube placement for otitis media. In this observational study, results of OtoSight imaging will not affect patient standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Children (17 years old or younger) scheduled for tympanostomy tube placement

Exclusion Criteria:

* Otoscopy contra-indicated or not possible per attending physician's decision

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children diagnosed with otitis media and scheduled for tympanostomy tube surgery.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
OtoSight imaging exam | 1-5 minutes
  Optical coherence tomography imaging to evaluate the middle ear.

SECONDARY OUTCOMES:
Adverse events | Date of recruitment (day of surgery) to post-operative follow-up visit (approx. 1 month, but can be longer)
  Rate of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Shelton, PhD, Principal Investigator — PhotoniCare, Inc.
Locations (2):
- United States (2):
  - Children's National Health System, Washington D.C., District of Columbia
  - Carle Foundation Hospital, Urbana, Illinois

IPD SHARING:
Plan to Share IPD: No